CLINICAL TRIAL: NCT02543151
Title: Prospective Evaluation of SpyGlass Direct Visualization System in Post Liver Transplant Biliary Stricture.
Brief Title: SpyGlass in Post Liver Transplant Biliary Complications.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Israelita Albert Einstein (Other)
Responsible Party: Principal Investigator, FERNANDA PRATA MARTINS, Attending physician, Hospital Israelita Albert Einstein
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1439-11; 28005314.5.0000.0071 (Other: CONEP)
Record Dates: First submitted 2015-09-02; First posted 2015-09-07 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Liver Transplant Disorder; Biliary Anastomosis Complication
Keywords: Biliary stricture; Cholangioscopy; Spyglass; Liver transplant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SpyGlass Choledochoscopy procedure (Experimental): Any patient referred to endoscopic management for biliary post liver transplant complication without previous treatment will be submitted to SpyGlass (direct visualization system) choledochoscopy procedure.
  Interventions: Procedure: SpyGlass (direct visualization system) choledochoscopy

INTERVENTIONS:
Procedure: SpyGlass (direct visualization system) choledochoscopy — SpyGlass (direct visualization system) choledochoscopy procedure will be performed pre and post biliary complication treatment

SUMMARY:
The purpose of this study is to describe SpyGlass choledochoscopy in patients with post orthotopic liver transplant (OLT) biliary strictures prior to endoscopic therapy and ductal changes after treatment stents.

DETAILED DESCRIPTION:
A prospective observational clinical study to be conducted in Hospital Israelita Albert Einstein, a large open-access, private tertiary referral center.

Consecutive eligible patients with suspected post OLT biliary complications referred to endoscopic retrograde cholangiopancreatography (ERCP) will be considered to SpyGlass as follows.

In those patients with confirmed biliary stricture, SpyGlass direct choledochoscopy will be performed prior to endoscopic treatment with stents.

After final stent removal, choledochoscopy will be repeated to evaluate biliary ductal mucosa.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred to endoscopic management for biliary post liver transplant complication without previous treatment

Exclusion Criteria:

* Patients referred to endoscopic management for biliary post liver transplant complication with any previous treatment.
* Below 18 years of age
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Documentation of biliary ductal changes in post-liver transplant biliary complications. | 2 years
  The study aim is to describe biliary ductal changes in post-liver transplant presenting biliary complications

SECONDARY OUTCOMES:
Number of Participants with Adverse Events. | 2 years
  Secondary outcomes include the description of adverse events

OTHER OUTCOMES:
Procedural success rate: | 1 year
  defined as the proportion of SpyGlass procedures completed where the diagnostic or therapeutic objectives were achieved.

CONTACTS AND LOCATIONS:
Overall Officials: ANGELO P FERRARI, MD, Study Director — Attending physician; FERNANDA P MARTINS, MD, Principal Investigator — Attending physician
Locations (1):
- Hospital Israelita Albert Einstein, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chen YK, Pleskow DK. SpyGlass single-operator peroral cholangiopancreatoscopy system for the diagnosis and therapy of bile-duct disorders: a clinical feasibility study (with video). Gastrointest Endosc. 2007 May;65(6):832-41. doi: 10.1016/j.gie.2007.01.025. PMID 17466202
- [Background] Draganov PV, Lin T, Chauhan S, Wagh MS, Hou W, Forsmark CE. Prospective evaluation of the clinical utility of ERCP-guided cholangiopancreatoscopy with a new direct visualization system. Gastrointest Endosc. 2011 May;73(5):971-9. doi: 10.1016/j.gie.2011.01.003. Epub 2011 Mar 17. PMID 21419408
- [Background] Tringali A, Lemmers A, Meves V, Terheggen G, Pohl J, Manfredi G, Hafner M, Costamagna G, Deviere J, Neuhaus H, Caillol F, Giovannini M, Hassan C, Dumonceau JM. Intraductal biliopancreatic imaging: European Society of Gastrointestinal Endoscopy (ESGE) technology review. Endoscopy. 2015 Aug;47(8):739-53. doi: 10.1055/s-0034-1392584. Epub 2015 Jul 6. PMID 26147492
- [Background] Hasan M, Canipe A, Tharian B, Navaneethan U, Varadarajulu S, Hawes R. Digital cholangioscopy-directed removal of a surgical staple from a strictured bile duct. Gastrointest Endosc. 2015 Nov;82(5):958. doi: 10.1016/j.gie.2015.05.035. Epub 2015 Jun 25. No abstract available. PMID 26117180